CLINICAL TRIAL: NCT01419665
Title: A Randomized, Controlled, Double-Blind Phase III Trial to Compare the Efficacy, Safety and Pharmacokinetics of GP2013 vs. MabThera® in Patients With Previously Untreated, Advanced Stage Follicular Lymphoma
Brief Title: GP2013 in the Treatment of Patients With Previously Untreated, Advanced Stage Follicular Lymphoma (ASSIST_FL)
Acronym: ASSIST_FL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP13-301; 2010-019522-13 (EudraCT Number); NCT03814785 (obsolete NCT alias)
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; Biosimilar; GP13-301; rituximab; Antibodies; CD20
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: A subset of patients is switched from GP2013 to MabThera or continued with MabThera during the maintenance phase, for these patients the treatment is finished as an open labeled parallel arm study. The original treatment assignment is kept blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP2013 (Experimental): Type: Biological/Vaccine
  Interventions: Biological: GP2013
- rituximab (Active Comparator): Type: Biological/Vaccine
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: GP2013 — Type: Biological/Vaccine
  Other Names: no brand name available
  Arms: GP2013
Biological: rituximab — Type: Biological/Vaccine
  Other Names: MabThera(R)
  Arms: rituximab

SUMMARY:
The purpose of this study is to demonstrate comparability of the ORR in patients with previously untreated, advanced stage FL who receive GP2013-treatment to patients who receive MabThera-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with previously untreated advanced stage, CD20-positive FL
* Patient with ECOG performance status 0, 1 or 2.

Exclusion Criteria:

* Patient with Grade 3b (aggressive) FL or any histology other than FL grade 1, 2 or 3a
* Patient who has previously received any prior therapy for lymphoma
* Patient with evidence of any uncontrolled, active infection (viral, bacterial or fungal).
* Patient with any malignancy within 5 years prior to date of randomization, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2015-07-10 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (153):
- Argentina (3):
  - Investigative site, La Plata
  - Investigative site, Rosario
  - Investigative site, San Miguel de Tucumán
- Australia (5):
  - Investigative site, Adelaide
  - Investigative site, Ballarat
  - Investigative site, Epping
  - Investigative site, Footscray
  - Investigative site, Wodonga
- Austria (2):
  - Investigative site, Graz
  - Investigative site, Vienna
- Brazil (15):
  - Investigative site, Barretos
  - Investigator site, Barretos
  - Investigative site, Botucatu
  - Investigative site, Campinas
  - Investigative site, Curitiba
  - Investigative site, Florianópolis
  - Investigative site, Fortaleza
  - Investigative site, Goiânia
  - Investigative site, Jaú
  - Investigative site, Passo Fundo
  - Investigative site, Porto Alegre
  - Investigative Site, Rio de Janeiro
  - Investigative site, Santo André
  - Investigative site, São Paulo
  - Investigative site, Sorocaba
- Bulgaria (5):
  - Investigative site, Pleven
  - Investigative site, Plovdiv
  - Investigative site, Rousse
  - Investigative site, Sofia
  - Investigative site, Varna
- Colombia (2):
  - Investigative site, Medellín
  - Investigative site, Montería
- France (3):
  - Investigative site, Colmar
  - Investigative site, Nîmes
  - Investigative site, Strasbourg
- Germany (2):
  - Investigative site, Bad Saarow
  - Investigative site, Koblenz
- Greece (4):
  - Investigative site, Athens
  - Investigative site, Ioannina
  - Investigative site, Larissa
  - Investigative site, Pátrai
- Hungary (2):
  - Investigative site, Győr
  - Investigative site, Kaposvár
- India (16):
  - Investigative site, Ahmedabad
  - India, Amritsar
  - Investigative site, Aurangabad
  - Investigative site, Bangalore
  - Investigative site, Chennai
  - Investigative site, Hyderabad
  - Investigative site, Kolkata
  - Investigtive site, Kolkata
  - Investigative site, Madurai
  - Investigative site, Mumbai
  - Investigative site, Nashik
  - Investigative site, New Delhi
  - Investigative site, Pune
  - Investigative site, Surat
  - Investigative site, Trivandrum
  - Investigative site, Vellore
- Ireland (3):
  - Investigative site, Dublin
  - Investigative site, Limerick
  - Investigative site, Waterford
- Israel (2):
  - Investigative site, Ashkelon
  - Investigative site, Nahariya
- Italy (11):
  - Investigative site, Bari
  - Investigative site, Florence
  - Investigative site, Meldola
  - Investigative site, Milan
  - Investigative site, Palermo
  - Investigative site, Pavia
  - Investigative site, Pescara
  - Investigative site, Piacenza
  - Investigative site, Ravenna
  - Investigative site, Reggio Calabria
  - Investigative site, Varese
- Japan (14):
  - Investigative site, Aomori
  - Investigative site, Fukuoka
  - Investigative site, Gifu
  - Investigative site, Kagoshima
  - Investigative site, Kitakyushu
  - Investigative site, Kobe
  - Investigative site, Komaki
  - Investigative site, Matsuyama
  - Investigative site, Okayama
  - Investigative site, Ōgaki
  - Invstigative site, Ōmura
  - Investigative site, Ōtake
  - Investigative site, Saga
  - Investigative site, Tachikawa
- Malaysia (11):
  - Investigative site, Alor Star
  - Investigative site, Ampang
  - Investigative site, George Town
  - Investigative site, Ipoh
  - Investigative site, Johor Bahru
  - Investigative site, Klang
  - Investigative site, Kuala Lumpur
  - Investigative site, Kuching
  - Investigative site, Malacca
  - Investigative site, Pulau Pinang
  - Investigative site, Subang Jaya
- Netherlands (8):
  - Investigative site, Amsterdam
  - Investigative site, Delft
  - Investigative site, Gouda
  - Investigative site, Heerlen
  - Investigative site, Rotterdam
  - Investigative site, Schiedam
  - Investigative site, Sittard
  - Investigative site, Zwolle
- Investigative site, Lima, Peru
- Poland (6):
  - Investigative site, Brzozów
  - Investigative site, Bydgoszcz
  - Investigative site, Chorzów
  - Investigative site, Krakow
  - Investigative site, Lublin
  - Investigative site, Warsaw
- Portugal (4):
  - Investigative site, Braga
  - Investigative site, Coimbra
  - Investigative site, Lisbon
  - Investigative site, Porto
- Romania (5):
  - Investigative site, Brasov
  - Investigative site, Bucharest
  - Investigative site, Cluj-Napoca
  - Investigative site, Iași
  - Investigative site, Timișoara
- Russia (8):
  - Investigative site, Arkhangelsk
  - Investigative site, Chelyabinsk
  - Investigative site, Krasnodar
  - Investigative site, Kursk
  - Investigative site, Moscow
  - Investigative site, Nizhny Novgorod
  - Investigative site, Rostov-on-Don
  - Investigative site, Saint Petersburg
- South Africa (5):
  - Investigative site, Cape Town
  - Investigative site, George
  - Investigative site, Johannesburg
  - Investigative site, Port Elizabeth
  - Investigative site, Pretoria
- Spain (6):
  - Investigative site, Barcelona
  - Investigative site, Donostia / San Sebastian
  - Investigative site, Madrid
  - Investigative site, Oviedo
  - Investigative site, Seville
  - Investigative site, Zaragoza
- Ukraine (7):
  - Investigative site, Cherkasy
  - Investigative site, Dnipropetrovsk
  - Investigative site, Donetsk
  - Investigative site, Ivano-Frankivsk
  - Investigative site, Kharkiv
  - Investigative site, Kyiv
  - Investigative site, Lviv
- United Kingdom (3):
  - Investigative site, Eastbourne
  - Investigative site, London
  - Investigative site, Worthing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jurczak W, Moreira I, Kanakasetty GB, Munhoz E, Echeveste MA, Giri P, Castro N, Pereira J, Akria L, Alexeev S, Osmanov E, Zhu P, Alexandrova S, Zubel A, Harlin O, Amersdorffer J. Rituximab biosimilar and reference rituximab in patients with previously untreated advanced follicular lymphoma (ASSIST-FL): primary results from a confirmatory phase 3, double-blind, randomised, controlled study. Lancet Haematol. 2017 Aug;4(8):e350-e361. doi: 10.1016/S2352-3026(17)30106-0. Epub 2017 Jul 14. PMID 28712941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 629 patients were randomized at 159 centers in 26 countries, 314 patients to GP2013 (312 patients treated) and 315 to MabThera. Of those 314 patients in the GP2013 group, 2 patients were randomized by error and discontinued before any treatment with GP2013. The number of patients in both treatment groups remained similar.
Pre-assignment Details: full analysis set participants : GP2013 312 MabThera 315 safety set participants : GP2013 312 MabThera 315 per protocol set participants: GP2013 310 MabThera 312 pharmacokinetic analysis set 1 : GP2013 119 MabThera 120 immunogenicity analysis set: GP2013 275 MabThera 287 pharmacodynamic analysis set : GP2013 24 MabThera 24
Groups:
- GP2013: Experimental Type: Biological/Vaccine
- Rituximab: Comparator Type: Biological/Vaccine
Period: Combination Treatment
Arm/Group | GP2013 | Rituximab
Started | 312 | 315
Completed (completed treatment at week 24) | 274 | 274
Not Completed | 38 | 41
Not completed — Adverse Event | 7 | 10
Not completed — Physician Decision | 5 | 8
Not completed — Protocol Violation | 6 | 2
Not completed — disease progression | 10 | 9
Not completed — Death | 5 | 7
Not completed — administrative problems | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4
Period: Maintenance Treatment and/or Follow up
Arm/Group | GP2013 | Rituximab
Started | 254 | 252
Completed | 132 | 150
Not Completed | 122 | 102
Not completed — switch to open label | 44 | 39
Not completed — administrative problems | 0 | 6
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 5 | 2
Not completed — disease progression | 53 | 37
Not completed — Death | 1 | 2
Not completed — Adverse Event | 11 | 7
Not completed — Lost to Follow-up | 1 | 2
Period: Open Label Phase
Arm/Group | GP2013 | Rituximab
Started | 44 | 39
Completed | 43 | 38
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — disease progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2013 | Rituximab | Total
Number analyzed (Participants) | 312 | 315 | 627
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.86) | 56.4 (11.72) | 56.9 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 169 | 350
  Male | 131 | 146 | 277
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian | 71 | 85 | 156
    Black | 6 | 3 | 9
    Caucasian | 214 | 207 | 421
    Native American | 2 | 5 | 7
    Other | 19 | 15 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Chinese | 5 | 6 | 11
    Hispanic / Latino | 59 | 68 | 127
    Indian (Indian Subcontinent) | 40 | 54 | 94
    Mixed Ethnicity | 8 | 3 | 11
    Other | 183 | 170 | 353
    Unknown / missing | 1 | 0 | 1
    Japanese | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of patients whose best overall disease response was either CR or PR during the combination treatment period based on blinded independent central radiology review.
Time Frame: 24 weeks
Population: per protocol set, participants with measure
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 311 | 313
percentage | 87.1 [83.59 to 90.15] | 87.5 [84.04 to 90.49]
Statistical Analysis 1: Comparison: GP2013 vs Rituximab; Test type: Equivalence — The equivalence margin of + or - 12% was determined considering the variability of the point estimate of the add-on effect by taking a value lower than the lower boundary of the 95% CI for Rituximab+chemotherapy versus chemotherapy obtained from historical data; Binomial approximation; difference in overall response rate = -0.40, 95% CI 2-sided [-5.94 to 5.14]

2. Secondary Outcome: To Evaluate the Complete Response (CR) Rate During the Combination Treatment Period
Time Frame: 24 weeks
Population: per protocol set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 311 | 313
Participants | 46 | 42

3. Secondary Outcome: To Evaluate the Partial Response (PR) Rate During the Combination Treatment Period
Time Frame: 24 weeks
Population: per protocol set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 311 | 313
Participants | 225 | 232

4. Secondary Outcome: To Evaluate the Progression Free Survival (PFS) With up to 3 Years of Follow-up Post Randomization
Description: Number of participants with progression free survival events
Time Frame: 3 years
Population: per protocol set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 312 | 315
Participants | 97 | 78
Statistical Analysis 1: Comparison: GP2013 vs Rituximab; Test type: Other — descriptive purposes, not powered for hypothesis testing; Regression, Cox; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.97 to 1.76]

5. Secondary Outcome: To Evaluate the Overall Survival (OS) With up to 3 Years of Follow-up Post Randomization, as Assessed by the Number of Deaths
Description: OS was defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died, OS was censored at the date of last contact including survival follow-up.
Time Frame: 3 years
Population: per protocol set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 312 | 315
Participants | 29 | 31
Statistical Analysis 1: Comparison: GP2013 vs Rituximab; Test type: Other — descriptive purposes, not powered for hypothesis testing; Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.55 to 1.52]

6. Secondary Outcome: To Evaluate the Incidence of Immunogenicity (ADA Formation) Against GP2013 and MabThera (Rituximab)
Description: number of participants with confirmed positive ADA
Time Frame: 24 weeks, 3 years
Population: immunogenicity set, participants with measure
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 275 | 287
Participants
  end of treatment combination phase (24 weeks): number analyzed (Participants) | 257 | 269
  end of treatment combination phase (24 weeks) | 1 | 2
  end of treatment manintenance phase (3 years): number analyzed (Participants) | 203 | 210
  end of treatment manintenance phase (3 years) | 1 | 0

7. Secondary Outcome: To Evaluate a PK Marker Following the Treatment With GP2013-Chemotherapy and MabThera-Chemotherapy (C Max)
Description: C max
  For descriptive purposes only, no hypothesis testing
Time Frame: day 63
Population: pharmacokinetic analysis set 1, participants with measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microg/mL
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 119 | 120
microg/mL | 333.59 (41.09) | 331.93 (35.32)

8. Secondary Outcome: To Evaluate a PK Marker Following the Treatment With GP2013-Chemotherapy and MabThera-Chemotherapy (C Trough)
Description: C through
  For descriptive purposes only, no hypothesis testing
Time Frame: day 63
Population: pharmacokinetic analysis set 1, participants with measure
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 119 | 120
microg/mL | 66.42 (47.593) | 82.13 (61.526)

9. Secondary Outcome: To Evaluate a PD Marker (Peripheral CD19+ B-cell Counts) Following the Treatment With GP2013 + Chemotherapy Amd MabThera- Chemotherapy
Description: AUEC (0-21d)
  For descriptive purposes only, no hypothesis testing
Time Frame: 21 days
Population: Pharmnacodynamic analysis set, participants with measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: %*day
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 24 | 24
%*day | 1790 (23.5) | 1910 (13.3)

10. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from the start of treatment up to 30 days after study drug discontinuation, for a maximum duration of 30 months (treatment duration ranged from 90 to 782 days) Deaths post treatment survival follow up were collected after the on- treatment period, up to 3 years.
Time Frame: 30 months, 3 years
Population: clinical data base population - treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituximab
Number analyzed (Participants) | 312 | 315
Participants
  on treatment death | 4 | 5
  on treatment deaths maintenance: number analyzed (Participants) | 254 | 252
  on treatment deaths maintenance | 2 | 2
  all deaths | 29 | 31

ADVERSE EVENTS:
Time Frame: On treatment AE, SAE and deaths were collected from the start of treatment up to 30/90 days after study drug discontinuation (30 days for combination phase and 90 for maintenance/open label phase), for a maximum duration of 30 months (treatment duration ranged from 90 to 782 days)
Description: Safety follow-up (treatment emergent AE/SAEs): after discontinuation of study treatment, all subjects were followed for safety for 30 days for combination phase and 90 for maintenance/open label phase.
Groups:
- Combination GP2013+CVP: Combination GP2013+CVP
- Combination MabThera+CVP: Combination MabThera+CVP
- Maintenance GP2013: Maintenance GP2013
- Maintenance MabThera: Maintenance MabThera
Arm/Group | Combination GP2013+CVP | Combination MabThera+CVP | Maintenance GP2013 | Maintenance MabThera
All-Cause Mortality (participants affected / at risk) | 4/312 | 5/315 | 2/254 | 2/252
Serious Adverse Events (participants affected / at risk) | 71/312 | 63/315 | 24/254 | 21/252
Other Adverse Events (participants affected / at risk) | 262/312 | 255/315 | 141/254 | 144/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination GP2013+CVP (N=312) | Combination MabThera+CVP (N=315) | Maintenance GP2013 (N=254) | Maintenance MabThera (N=252)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 9 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Polycystic liver disease (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 7 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4 | 3 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Sepsis (Infections and infestations) | 2 | 5 | 1 | 0
Septic shock (Infections and infestations) | 3 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0
Cervical cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 2 | 0
Meningeal disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination GP2013+CVP (N=312) | Combination MabThera+CVP (N=315) | Maintenance GP2013 (N=254) | Maintenance MabThera (N=252)
Anaemia (Blood and lymphatic system disorders) | 25 | 28 | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 23 | 25 | 11 | 5
Neutropenia (Blood and lymphatic system disorders) | 78 | 91 | 32 | 16
Abdominal pain (Gastrointestinal disorders) | 28 | 35 | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 20 | 16 | 4 | 7
Constipation (Gastrointestinal disorders) | 69 | 64 | 8 | 10
Diarrhoea (Gastrointestinal disorders) | 39 | 33 | 11 | 18
Nausea (Gastrointestinal disorders) | 51 | 42 | 11 | 8
Vomiting (Gastrointestinal disorders) | 22 | 26 | 6 | 12
Asthenia (General disorders) | 30 | 31 | 12 | 11
Fatigue (General disorders) | 35 | 31 | 6 | 10
Oedema peripheral (General disorders) | 13 | 24 | 4 | 11
Pyrexia (General disorders) | 27 | 32 | 12 | 13
Influenza (Infections and infestations) | 16 | 7 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 22 | 22 | 12 | 17
Urinary tract infection (Infections and infestations) | 27 | 22 | 14 | 25
Viral upper respiratory tract infection (Infections and infestations) | 8 | 10 | 5 | 15
Infusion related reaction (Injury, poisoning and procedural complications) | 41 | 37 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 17 | 21 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 22 | 4 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 18 | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21 | 9 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 30 | 14 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 20 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 24 | 7 | 14
Dizziness (Nervous system disorders) | 18 | 12 | 5 | 2
Headache (Nervous system disorders) | 29 | 34 | 12 | 14
Neuropathy peripheral (Nervous system disorders) | 49 | 30 | 8 | 2
Paraesthesia (Nervous system disorders) | 24 | 44 | 7 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 26 | 23 | 6 | 5
Insomnia (Psychiatric disorders) | 15 | 19 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 37 | 33 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 26 | 1 | 1
Hypertension (Vascular disorders) | 22 | 15 | 12 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.